CLINICAL TRIAL: NCT00860561
Title: Faslodex Post Marketing Surveillance
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D6997L00018
Record Dates: First submitted 2009-03-11; First posted 2009-03-12 (Estimated); Last update posted 2014-10-10 (Estimated); Status verified 2014-10

CONDITIONS: Breast Cancer
Keywords: Efficacy profile; Safety profile; Faslodex
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Postmenopausal women with locally advanced or metastatic breast cancer who have failed 2 or more prior hormone therapies, or were intolerant to prior hormone therapy and have no endocrine therapeutic options.

SUMMARY:
This PMS aims to assess the efficacy, the safety and tolerability profile of Faslodex in everyday practice. Secondary objective of this PMS is to identify the frequency of serious adverse events or any unknown adverse events of Faslodex.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women
* Patients who have failed 2 or more prior hormone therapies (The prior hormone therapies should contain both antiestrogen and non-steroidal Aromatase inhibitor)
* Patients who were intolerant to prior hormone therapy and have no endocrine therapeutic options (The prior hormone therapies should contain both antiestrogen and non-steroidal Aromatase inhibitor)

Exclusion Criteria:

* The patients who received Faslodex treatment before

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Postmenopausal women with locally advanced or metastatic breast cancer who have failed 2 or more prior hormone therapies, or were intolerant to prior hormone therapy and have no endocrine therapeutic options.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2009-01; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Adverse events are confirmed by investigator through asking to patients or patients' voluntary reporting. | 5 years
Efficacy of Faslodex is assessed by proper method among CT scan, MRI, Ultrasound, etc. The RECIST criteria for target and non-target lesions will be used to evaluate efficacy. | 5 years

CONTACTS AND LOCATIONS:
Locations (7):
- South Korea (7):
  - Research Site, Cheonan
  - Research Site, Daegu
  - Research Site, Daejeon
  - Research Site, Iksan
  - Research Site, Jeonju
  - Research Site, Seoul
  - Research Site, Suwon

REFERENCES:
- See also: CSR_Synopsis_D6997L00018 — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=592&filename=CSR_Synopsis_D6997L00018.pdf